CLINICAL TRIAL: NCT02003820
Title: Using Video Modeled Social Stories to Improve Oral Hygiene in Children With Autism
Brief Title: Using Video Modeled Social Stories to Improve Oral Hygiene in Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Ben Popple, Resident, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pedidentalautism
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Autism Spectrum Disorder; Dental Caries
Keywords: Autism; Dental Caries; Prevention; Oral Hygiene
MeSH Terms: conditions — Autism Spectrum Disorder; Dental Caries; Autistic Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Group 1 will receive plaque index exam and immediately start their three week intervention of watching a dental hygiene video immediately before brushing twice per day. Plaque index exams will be completed at start, t-10 days, and t-21 days. Parental surveys will be completed at each plaque index exam and 6 weeks after start.
  Interventions: Behavioral: video modeled social story
- Group 2 (Experimental): Group 2 will receive plaque index exam and immediately start their three week intervention of watching a control video immediately before brushing twice per day. Plaque index exams will be completed at start, t-10 days, and t-21 days. Parental surveys will be completed at each plaque index exam and 6 weeks after start.
  Interventions: Behavioral: video modeled social story

INTERVENTIONS:
Behavioral: video modeled social story — Patient will watch a Youtube compatible video of a child in the same age range as the study participants demonstrating proper brushing technique. The video will be paired with written subtitles created using the Social Story format. The subtitles will be read to the participant as the video plays. The patient will watch the video immediately before each brushing session morning and night for the three week intervention. After the intervention period the video will be made available on Youtube.com for the participants to use as they wish.

SUMMARY:
We hypothesize that oral hygiene habits in children 8-12 years of age can be improved using video format Social Story intervention techniques. The purpose of this study is to investigate the effectiveness of video format social stories used to inform and educate children and parents about proper dental hygiene technique over a 6 week intervention period. We will measure the success of intervention using data collected from clinical exams and caregiver/participant surveys. Evaluation of data collected will be used to determine the effectiveness of the intervention.

DETAILED DESCRIPTION:
In this pilot study improvement of tooth brushing practices in children with Autism Spectrum Disorder between the ages of eight and twelve years old will be evaluated. Participants placed in two randomized groups will watch a Youtube format instructional video twice each day immediately before each brushing during the three-week intervention period.

The video intervention will teach participants to use the usual and customary hygiene skills. Participants will view a child in their age range demonstrating proper brushing using the Bass brushing technique. The video will also have written narration at the bottom of the screen delivering printed information using Social Story style prompts. The Social Story prompts will also be read aloud for auditory delivery of information. The video will be two to three minutes long.

Success of intervention will be determined using data collected at multiple times during the pilot. First, clinical exams will be completed before the intervention, half way through the intervention, and at the end of three weeks to evaluate how clean the patients oral cavity appears. Exams should take no more than twenty minutes in the dental chair. Second, Qualtrics emails will be sent to the patient's caregiver at 5:30 AM and 4:30 PM each day during intervention providing access to the instructional video. After opening the email and watching the video, there will be a simple "yes or no" survey question asking the caregiver if the video was watching before that brushing session. Finally, more in depth caregiver surveys will be completed at the end of each week during the intervention consisting of no more than fifteen questions. The surveys will evaluate the caregiver's perception of intervention success. At completion of the intervention the video will be made available to all participants via Youtube.com. One final survey will be sent to caregivers three weeks post intervention to determine if the video is still being used for hygiene reinforcement.

Multiple efforts for study control will be implemented. To control for the impact that watching a video twice a day may have Group 2 will watch a control video. Group 1 will watch a dental hygiene video. Clinical evaluators will also be blinded to prevent bias when evaluating the two groups clinically. One examiner will conduct initial exams. A second examiner will conduct all subsequent exams with no knowledge of what group each patient is assigned. Evaluators will be calibrated pre-study evaluating hygiene patients at the dental clinic.

All participants in this study will also be enrolled at Yale Child Study Center to measure the participants IQ using autism specific IQ testing methods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Autism Spectrum Disorder
* Access to internet and email at home
* Patient of record at Yale New Haven Hospital Pediatric Dental Clinic

Exclusion Criteria:

* Outside of specified age range
* No home access to email and internet

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Measure of video intervention use | 3 weeks
  Video intervention will be emailed to participants twice daily during intervention period. After watching video the patient will be given a one question survey asking if they watched the video before that brushing period.
Plaque index | 3 weeks
  Patients will be given a usual and customary dental exam in the clinic before intervention is introduced to evaluate level of oral hygiene by a blinded evaluator. Plaque index will also be measured in the usual and customary manor half way through intervention and at the end of intervention period.

SECONDARY OUTCOMES:
Caregiver survey | 6 weeks
  Caregivers will be given 10-15 question surveys at beginning of intervention, at the each week clinical visit during the intervention, and 3 weeks post intervention measuring their perception of the intervention's effect on the study subject. Questions will measure ease of completing brushing, perceived brushing effectiveness, amount of help patient requires to brush effectively, interest in video...

CONTACTS AND LOCATIONS:
Overall Officials: Ben S Popple, DMD, Principal Investigator — Yale Pediatric Dentistry; Fred Shic, PhD, Study Chair — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Hospital Pediatric Dental Center, New Haven, Connecticut
  - Yale Pediatric Dental Center Suite 403, New Haven, Connecticut

REFERENCES:
- [Background] Friedlander AH, Yagiela JA, Paterno VI, Mahler ME. The neuropathology, medical management and dental implications of autism. J Am Dent Assoc. 2006 Nov;137(11):1517-27. doi: 10.14219/jada.archive.2006.0086. PMID 17082277
- [Background] Volkmar, F.W., L,, A Practical Guide to Autism: what every parent, family member, and teacher needs to know. 2009, Hoboken, NJ: John Wiley & Sons, Inc. 610.
- [Background] Rice C, Schendel D, Cunniff C, Doernberg N. Public health monitoring of developmental disabilities with a focus on the autism spectrum disorders. Am J Med Genet C Semin Med Genet. 2004 Feb 15;125C(1):22-7. doi: 10.1002/ajmg.c.30006. PMID 14755430
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Text Revision (DSM-IVTR). 2000, Washington, DC: American Psychiatric Publishing.
- [Background] Marshall J, Sheller B, Mancl L. Caries-risk assessment and caries status of children with autism. Pediatr Dent. 2010 Jan-Feb;32(1):69-75. PMID 20298657
- [Background] Jaber MA. Dental caries experience, oral health status and treatment needs of dental patients with autism. J Appl Oral Sci. 2011 May-Jun;19(3):212-7. doi: 10.1590/s1678-77572011000300006. PMID 21625735
- [Background] Klein U, Nowak AJ. Characteristics of patients with autistic disorder (AD) presenting for dental treatment: a survey and chart review. Spec Care Dentist. 1999 Sep-Oct;19(5):200-7. doi: 10.1111/j.1754-4505.1999.tb01386.x. PMID 10765886
- [Background] Affairs, C.o.C., Guidelines on Caries-risk Assessment and Management for Infants, Children, and Adolescents. American Academy of Pediatric Dentistry Reference Manual, 2013. 35(6): p. 118-125.
- [Background] Capozza LE, Bimstein E. Preferences of parents of children with autism spectrum disorders concerning oral health and dental treatment. Pediatr Dent. 2012 Nov-Dec;34(7):480-4. PMID 23265165
- [Background] DeMattei R, Cuvo A, Maurizio S. Oral assessment of children with an autism spectrum disorder. J Dent Hyg. 2007 Summer;81(3):65. Epub 2007 Jul 1. PMID 17908421
- [Background] Rada RE. Controversial issues in treating the dental patient with autism. J Am Dent Assoc. 2010 Aug;141(8):947-53. doi: 10.14219/jada.archive.2010.0308. PMID 20675420
- [Background] Loo CY, Graham RM, Hughes CV. The caries experience and behavior of dental patients with autism spectrum disorder. J Am Dent Assoc. 2008 Nov;139(11):1518-24. doi: 10.14219/jada.archive.2008.0078. PMID 18978390
- [Background] Marshall J, Sheller B, Mancl L, Williams BJ. Parental attitudes regarding behavior guidance of dental patients with autism. Pediatr Dent. 2008 Sep-Oct;30(5):400-7. PMID 18942599
- [Background] Stein LI, Polido JC, Najera SO, Cermak SA. Oral care experiences and challenges in children with autism spectrum disorders. Pediatr Dent. 2012 Sep-Oct;34(5):387-91. PMID 23211914
- [Background] Weil TN, Inglehart MR. Three- to 21-year-old patients with autism spectrum disorders: parents' perceptions of severity of symptoms, oral health, and oral health-related behavior. Pediatr Dent. 2012 Nov-Dec;34(7):473-9. PMID 23265164
- [Background] Orellana LM, Martinez-Sanchis S, Silvestre FJ. Training adults and children with an autism spectrum disorder to be compliant with a clinical dental assessment using a TEACCH-based approach. J Autism Dev Disord. 2014 Apr;44(4):776-85. doi: 10.1007/s10803-013-1930-8. PMID 24002415
- [Background] Cardon TA, Wilcox MJ. Promoting imitation in young children with autism: a comparison of reciprocal imitation training and video modeling. J Autism Dev Disord. 2011 May;41(5):654-66. doi: 10.1007/s10803-010-1086-8. PMID 20697791
- [Background] Charlop MH, Milstein JP. Teaching autistic children conversational speech using video modeling. J Appl Behav Anal. 1989 Fall;22(3):275-85. doi: 10.1901/jaba.1989.22-275. PMID 2793634
- [Background] Bohlander AJ, Orlich F, Varley CK. Social skills training for children with autism. Pediatr Clin North Am. 2012 Feb;59(1):165-74, xii. doi: 10.1016/j.pcl.2011.10.001. PMID 22284800
- [Background] Litras S, Moore DW, Anderson A. Using video self-modelled social stories to teach social skills to a young child with autism. Autism Res Treat. 2010;2010:834979. doi: 10.1155/2010/834979. Epub 2010 Jun 9. PMID 22937239
- [Background] Karkhaneh M, Clark B, Ospina MB, Seida JC, Smith V, Hartling L. Social Stories to improve social skills in children with autism spectrum disorder: a systematic review. Autism. 2010 Nov;14(6):641-62. doi: 10.1177/1362361310373057. Epub 2010 Oct 5. PMID 20923896
- [Background] Kokina A, Kern L. Social Story interventions for students with autism spectrum disorders: a meta-analysis. J Autism Dev Disord. 2010 Jul;40(7):812-26. doi: 10.1007/s10803-009-0931-0. PMID 20054628
- [Background] Ali, S.F., N., Investigating the Evidence Base of Social Stories. Educational Psycology in Practice, 2006. 22(4): p. 355-377.